CLINICAL TRIAL: NCT03173859
Title: A Randomized Phase II Study to Investigate the Efficacy of Rotations Between Abiraterone Acetate and Apalutamide Versus Sequential Administration in Chemo-naïve Metastatic Castration Resistant Prostate Cancer Patients
Brief Title: Efficacy of Rotations Between Abiraterone Acetate and Apalutamide in mCRPC Patients
Acronym: AERA
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Delayed initiation
Sponsor: University of Athens (Other)
Responsible Party: Principal Investigator, Aristotelis Bamias, Professor, University of Athens
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 70/3/14073; 2017-000443-41 (EudraCT Number)
Record Dates: First submitted 2017-05-28; First posted 2017-06-02 (Actual); Last update posted 2020-11-18 (Actual); Status verified 2020-11

CONDITIONS: Prostatic Neoplasms, Castration-Resistant
Keywords: prostate cancer, abiraterone, apalutamide
MeSH Terms: conditions — Prostatic Neoplasms, Castration-Resistant; Prostatic Neoplasms | interventions — abiraterone; Abiraterone Acetate; apalutamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Rotational (Experimental): Abiraterone acetate 1000mg qD and prednisone 5mg bid administered orally starting on Day 1 of Cycle 1 for 3 cycles, followed by apalutamide 240mg qD orally for 3 cycles. The duration of each cycle is 28 days
  Interventions: Drug: Abiraterone; Drug: Apalutamide
- Sequential (Active Comparator): Abiraterone acetate 1000mg qD and prednisone 5mg bid administered orally starting on Day 1 of Cycle 1 until disease progression, followed by apalutamide 240mg qD orally until second disease progression.
  Interventions: Drug: Abiraterone; Drug: Apalutamide

INTERVENTIONS:
Drug: Abiraterone — Abiraterone acetate 1000mg qD and prednisone 5mg bid administered orally
  Other Names: Zytiga
Drug: Apalutamide — apalutamide 240mg qD orally

SUMMARY:
A randomized phase II study comparing the sequential use of abiraterone followed after progression by apalutamide with alternating cycles of abiraterone and apalutamide

DETAILED DESCRIPTION:
This is an open-label, randomized phase II study to investigate the feasibility of alternating cycles of treatment with abiraterone plus prednisone and apalutamide compared to sequential treatment of abiratereone plus prednisone followed by apalutamide. 7 centers in Greece will participate in the study.

The study population consists of adult patients (over 18 years old) with histologically confirmed metastatic prostate adenocarcinoma who have disease progression - as defined by PCWG2 criteria - despite androgen deprivation therapy and who have not received prior therapy for their castration resistant disease.

The purpose of the study is to determine the progression free survival, feasibility and safety profile of the experimental arm compared to standard of care.

In the experimental arm alternating treatment will consist of repeating cycles of 24 weeks of treatment consisting of 12 weeks of abiraterone acetate 1000mg orally qd and prednisone 5mg orally bid, followed by 12 weeks of apalutamide 240 mg per day. There will be no wash out period between cycles.

The comparative arm will be the standard regimen of abiraterone 1000mg orally qd plus prednisone 5mg orally bid until progression, followed thereafter by apalutamide 240mg orally qd until progression.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Age >18 years Histologically confirmed metastatic or advanced prostate cancer adenocarcinoma that has received no treatment for the castration resistant disease and has progressed during treatment with complete androgen blockade (luteinizing hormone releasing hormone agonist or antagonist and an antiandrogen eg. Bicalutamide).

Availability of a representative formalin-fixed, paraffin-embedded tumor specimen (FFPE) that enabled definitive diagnosis of prostate cancer.

Two rising PSA levels >2ng/ml measured 1 week apart during or following the most recent prior therapy for prostate cancer (PCWG2 criteria) or radiographic evidence of disease progression in bone with or without biochemical disease progression on the basis of the PSA value.

Ongoing androgen deprivation, with serum testosterone <50ng/dl ECOG performance status 0-1 at screening Adequate hematologic and organ function within 14 days before the first study treatment (hematologic parameters must be assessed >14 days after a prior transfusion, if any) as defined by

* Hemoglobin >9g/dl
* Neutrophils >1500/μL
* Platelet count >100000/μL
* Total bilirubin <1,5xULN with the following exception:

  o Patients with known Gilbert syndrome who have serum bilirubin<3xULN
* AST and ALT<2,5xULN with the following exception

  o Patients with bone-only metastasis may have AST<5xULN, provided that ALT <2,5xULN and total bilirubin <1,5xULN
* Serum albumin >3g/dl
* Serum potassium ≥3.5mmol/L
* Serum creatinine <1,5xULN or creatinine clearance of >50ml/min based on Cockcroft-Gault equation
* Agreement by patient and/or partner to use an effective form of contraception including surgical sterilization, reliable barrier method, birth control pills, contraceptive hormone implants or true abstinence and to continue its use for the duration of the study and for 6 months after the last dose of study treatment.

Exclusion Criteria:

* Small cell or neuroendocrine prostate carcinoma Inability or unwillingness to swallow pills Malabsorption syndrome or other condition that would interfere with enteral absorption Congenital long QT syndrome or QTc>480msec NYHA Class II to IV heart failure or LVEF <50% or ventricular arrhythmia requiring medication Previous therapy for prostate cancer with CYP17 inhibitors including ketoconazole or investigational agents (VMT-VT-464, Orteronel etc) or novel antiandrogens (enzalutamide of OMD-208) for more than 7 days Presence of visceral metastasis History of another invasive cancer within 3 years from screening, with the exception of fully treated cancers with a remote probability of recurrence Duration of previous Androgen Deprivation Therapy <12months Active infection requiring IV antibiotics

Clinically significant cardiovascular disease including the following:

* unstable angina,
* myocardial infarction within 6 months from screening, or
* cerebrovascular accident within 6 months from screening Major surgical procedure within 4 weeks prior to initiation of study treatment Treatment with an investigational agent within 4 weeks prior to initiation of study treatment Unresolved, clinical significant toxicity from prior treatment Hypersensitivity reaction to the active pharmaceutical ingredient or any of the tablet components Any medical condition that restrain the patient to comply with study and follow-up procedures Inability to comply with study and follow up procedures

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-01 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Radiographic progression-free survival | Estimated up to 24 months
  time until radiographic progression as assessed by PCWG2 criteria

SECONDARY OUTCOMES:
Overall survival | estimated up to 36 months
  time until death or lost to follow up
Time to cytotoxic therapy initiation | Estimated up to 24 months
  time until the beginning of chemotherapy
Time until PSA progression | Estimated up to 24 months
  time until PSA progression as defined by PCWG2 criteria
Incidence, nature and severity of AEs | Estimated up to 24 months
  recording of all AE/SAEs

OTHER OUTCOMES:
Patient reported outcomes assessed using the FACT-P and EQ-5D-5L questionnaires | Estimated up to 24 months
  Differences in FACT-P questionnaires between treatment groups
Number of Circulating Tumor Cells (CTCs) and ARv7 analysis in CTCs from peripheral blood at baseline evaluation, first and second disease progression in Arm 2 and disease progression in Arm 1 (PD1). | Estimated up to 24 months
  Correlation of CTCs number and ARv7 expression with rPFS and OS in these patients
Patient reported outcomes assessed using the EQ-5D-5L questionnaires | Estimated up to 24 months
  Differences in EQ-5D-5L questionnaires between treatment groups

IPD SHARING:
Plan to Share IPD: No